CLINICAL TRIAL: NCT00130299
Title: An 18-month Randomized Controlled Trial of a Low Glycemic Load Diet
Brief Title: An 18-month Trial of a Low Glycemic Load Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Charles H. Hood Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59240-#1; R01DK059240 (NIH)
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Fat-Restricted

INTERVENTIONS:
Behavioral: low glycemic load diet
Behavioral: low fat diet

SUMMARY:
The primary aim of this study is to compare the effects of an experimental low-glycemic load diet with those of a conventional low-fat diet among obese young adults in an 18-month randomized-controlled trial.

DETAILED DESCRIPTION:
The prevalence of obesity has risen dramatically among children in the U.S. since the 1960s. Effective treatment of childhood obesity is widely recognized as instrumental to public health efforts to combat type 2 diabetes and heart disease. Evidence from animal studies, short-term human studies and epidemiology suggests that diets designed to minimize the rise in postprandial blood glucose, that is low glycemic index, may be useful in the treatment of obesity and related complications. This project proposes an month RCT comparing a low glycemic load diet to a conventional low fat diet. Both diet groups will receive identical treatment intensity, behavioral modification and physical activity recommendations. The primary endpoint will be change in percent body fat by dexa-scan at 18 months; other outcomes include insulin resistance and CVD risk factors. Compliance will be assessed by interviewer-administered, 24-hour dietary recalls.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35 years
* Body mass index (BMI) ≥ 30 kg/m2
* Access to a working telephone
* Conversant in English
* Written medical clearance from a primary care physician or nurse practitioner, ruling out any pre-existing or complicating medical condition

Exclusion Criteria:

* Body weight >300 lbs
* Major medical illness (heart, kidney or liver disease; diabetes; cancer; endocrinopathy; psychiatric illness) or other active medical problem
* An obesity-associated genetic syndrome (e.g., Prader-Willi)
* An abnormal screening laboratory test (ALT, creatinine, BUN, hematocrit)
* Fasting blood glucose ≥ 126 mg/dl)
* Taking any prescription medication that affects body weight (glucocorticoids, neuropsychiatric agents), blood pressure, or serum cholesterol concentrations
* Currently smoking (1 cigarette during any of the last 7 days)
* Previous diagnosis of an eating disorder (anorexia nervosa, bulimia, binge-eating disorder)
* If female, not pregnant or planning to become pregnant in the next 18 months and not lactating
* Failure to complete the pre-enrollment visits

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2004-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
change in adiposity as measured by dual energy x-ray absorptiometry (DEXA).

SECONDARY OUTCOMES:
change in insulin resistance as measured by the homeostasis model assessment; change in glucose tolerance as measured by an oral glucose tolerance test (OGTT); change in cardiovascular disease risk factors

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; Cara B Ebbeling, PhD, Study Director — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ebbeling CB, Leidig MM, Sinclair KB, Seger-Shippee LG, Feldman HA, Ludwig DS. Effects of an ad libitum low-glycemic load diet on cardiovascular disease risk factors in obese young adults. Am J Clin Nutr. 2005 May;81(5):976-82. doi: 10.1093/ajcn/81.5.976. PMID 15883418
- [Result] Ebbeling CB, Leidig MM, Feldman HA, Lovesky MM, Ludwig DS. Effects of a low-glycemic load vs low-fat diet in obese young adults: a randomized trial. JAMA. 2007 May 16;297(19):2092-102. doi: 10.1001/jama.297.19.2092. PMID 17507345